CLINICAL TRIAL: NCT06364202
Title: Effects of Peanut Butter on Sleep Quality and Daily Energy Levels in Fire Fighters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, Angelia Holland, Associate Professor, Augusta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1928368
Record Dates: First submitted 2024-04-09; First posted 2024-04-15 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Sleep; Body Composition; Blood Pressure; Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Did not receive peanut butter, maintained normal diet and activity. Asked to stop eating 2 hours prior to bed for 7 weeks.
- Peanut Butter (Experimental): Received and asked to consume 2 tbsp of peanut butter 2 hours before bedtime 5 nights per week for 7 weeks and to stop eating after that before bed. Other than that, asked to maintain normal diet and activity.
  Interventions: Dietary Supplement: Peanut Butter

INTERVENTIONS:
Dietary Supplement: Peanut Butter — 2 tablespoons of peanut butter
  Arms: Peanut Butter

SUMMARY:
The purpose of this study is to examine the possible benefits of peanut butter consumption prior to bedtime on sleep and energy levels among fire fighters. Fire fighters require high levels of energy to perform their occupational tasks but commonly lack sleep as well as the amount of dietary protein and fat suggested for tactical athletes. By addressing this gap, we expect that if peanut butter consumption is shown to improve sleep and/or energy, this lifestyle change (peanut butter consumption) may be appealing to fire fighters because of the ease and low cost of peanut butter. Aim 1: Determine if consuming peanut butter prior to bedtime alters measures of sleep quality and quantity in fire fighters. It is hypothesized that firefighters who consume the peanut butter will have positive impacts in measure of sleep quality and energy levels.

Aim 2: Examine the effects of peanut butter consumption on morning and evening energy levels

DETAILED DESCRIPTION:
This study will utilize a randomized, parallel-arm, placebo-controlled design to determine the impact peanut butter consumption may have on sleep and energy levels in firefighters when consumed before bed-time. Forty local fire fighters will be recruited to complete this eight-week study; week one will constitute a baseline and weeks 2-8 will consist of the intervention. A blinded statistician will randomize the participants into one of two groups: a control group and a peanut butter group. During the first familiarization visit, all participants will sign an informed consent, receive height and weight measurements, waist and hip circumference measurements, blood pressure measurement, fill out a 30-day diet recall, fill out 3 questionnaires (Insomnia Severity Index, PTSD-checklist 5 (PCL-5), and Dispositional Resilience; will take 10 minutes to fill out) and receive a validated sleep monitor (Actigraph GT3X watch and heart rate monitor chest strap) and 14 Visual Analogue Scale (VAS) questionnaires which assess energy levels and time of last caffeine, alcohol, and screen time before bed. They will wear the watch for seven days along with the heart rate monitor for 5 nights and complete the VAS twice a day for seven days on qualtrics while maintaining a normal diet and physical activity. A link to take the surveys will be provided during the familiarization visit. After this baseline week, participants will then continue to wear the Actigraph watch daily for seven weeks and fill out a VAS twice a day while taking part in their specified intervention. Those in the control group will proceed with the same protocol as for the baseline week. Those in the peanut butter group will also continue with the same protocol as in the baseline week with the addition of consuming two tablespoons of peanut butter two hours before bed for five nights a week during the seven-week intervention. We will provide a tablespoon measurer and three jars of natural peanut butter to the participants in the peanut butter group. To increase ease of participation, we will meet in a private room at the local fire stations to collect data. Both the peanut butter and control group will be asked not to eat anything two hours before bed during those five days (after the peanut butter serving in the peanut butter group). The peanut butter consumption is dependent on randomization group assignment. Participants in both groups will be asked to maintain their normal diet and not change their physical activity levels and/or begin a weight loss program throughout their time in the study (approximately eight-weeks).

ELIGIBILITY:
Inclusion Criteria:

* Works for local fire department, employed full-time

Exclusion Criteria:

* Under 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Body composition | Baseline
  BIA to assess body fat and lean body mass.
Body composition | Immediately after the intervention
  BIA to assess body fat and lean body mass.
Sleep | 8 weeks
  Assessed sleep throughout the study for 8 weeks via actigraph monitor
Blood pressure | Baseline
  Assessed blood pressure
Blood pressure | Immediately after the intervention
  Assessed blood pressure

SECONDARY OUTCOMES:
Physical activity | 8 weeks
  Assessed activity throughout the study for 8 weeks via actigraph monitor

CONTACTS AND LOCATIONS:
Locations (1):
- Augusta University, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided